CLINICAL TRIAL: NCT04033159
Title: A Phase 1/2 Trial on the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Exploratory Efficacy of DYN101 in Patients ≥ 16 Years of Age With Centronuclear Myopathies Caused by Mutations in DNM2 or MTM1.
Brief Title: Early Phase Human Drug Trial to Investigate Dynamin 101 (DYN101) in Patients ≥ 16 Years With Centronuclear Myopathies
Acronym: Unite-CNM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on tolerability findings at the low dose level thus far, continuation of dosing or even dose escalation is not possible.
Sponsor: Dynacure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DYN101-C101
Record Dates: First submitted 2019-06-12; First posted 2019-07-25 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Centronuclear Myopathy
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Intervention Model Description: Trial consisting of pre-screening consent, screening period, run-in period (if applicable), SAD part with 4 weeks follow-up after IMP and washout period of ≥ 12 weeks, MAD part of 12 weeks and MAD extension part of 12 weeks. All subjects to participate in SAD, MAD, and MAD extension unless they withdraw. Subjects to receive DYN101 in a low (1.5 mg/kg), middle (4.5 mg/kg) or high (9 mg/kg) dose in Cohorts 1, 2 and 3 respectively, and remain on assigned dose throughout the trial (unless IDMC advises otherwise). Each cohort will have 3-4 subjects with a DNM2 mutation and 2-3 subjects with a MTM1 mutation. Cohorts will enroll in a sequential staggered approach with an interval of ≥7 days between dosing of the first and the next subject in a cohort (after Medical Monitor 48hr safety data review).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- cohort 1 (Experimental): DYN101 in a low dose (1.5 mg/kg), (unless the independent data monitoring committee [IDMC] advises otherwise). In each cohort, there will be 3-4 subjects with a mutation in DNM2 (subcohort a) and 2-3 subjects with a mutation in MTM1 (subcohort b).
  Interventions: Drug: DYN101
- cohort 2 (Experimental): DYN101 in a middle dose (4.5 mg/kg), (unless the IDMC advises otherwise). In each cohort, there will be 3-4 subjects with a mutation in DNM2 (subcohort a) and 2-3 subjects with a mutation in MTM1 (subcohort b).
  Interventions: Drug: DYN101
- cohort 3 (Experimental): DYN101 in a high dose (9 mg/kg), (unless the IDMC advises otherwise). In each cohort, there will be 3-4 subjects with a mutation in DNM2 (subcohort a) and 2-3 subjects with a mutation in MTM1 (subcohort b).
  Interventions: Drug: DYN101

INTERVENTIONS:
Drug: DYN101 — DYN101, is a constrained ethyl gapmer ASO directed against human DNM2 RNA
  Other Names: there is no other intervention name

SUMMARY:
There are no available treatments aside from supportive care for patients with Centronuclear myopathy (CNM). This trial will assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD)/preliminary efficacy of a new medicine called DYN101 in patients ≥ 16 years of age with CNM caused by mutations in Dynamin2 (DNM2) or Myotubularin1 (MTM1).

The trial will consist of a consent, a screening period, a run-in period (if applicable), a Single dose treatment part (SAD) with 4 weeks of follow-up after the drug administration and a washout period of at least 12 weeks (followed by follow-up phone calls), a Multiple dose treatment part (MAD) of 12 weeks of weekly dosing, and a Multiple dose extension part of 12 weeks. All subjects will participate in the SAD, MAD, and MAD extension parts, unless they withdraw. During this time, multiple test will be performed in order to better understand how the drug is distributed and then later removed from the body and whether there any signs of an effect.

As this trial is investigational, there is no defined, expected benefit for subjects who participate in this trial except a better knowledge of their disease.

DETAILED DESCRIPTION:
There are currently no available treatments aside from supportive care for patients with Centronuclear myopathy (CNM). This trial will assess the safety, tolerability, PK and PD/preliminary efficacy of DYN101 in patients ≥ 16 years of age with CNM caused by mutations in DNM2 or MTM1.

DYN101 is a synthetically manufactured constrained ethyl gapmer antisense oligonucleotide (ASO) directed against DNM2 pre-messenger ribonucleic acid (mRNA). DYN101 will be provided as a sterile concentrated solution for reconstitution into an infusion solution for intravenous (IV) administration, and will be diluted into a 0.9% sodium chloride solution before administration.

The trial will consist of a pre-screening consent, a screening period, a run-in period (if applicable), a SAD part with 4 weeks of follow-up after investigational medicinal product (IMP) administration and a washout period of at least 12 weeks (followed by follow-up phone calls until the MAD part starts), a MAD part of 12 weeks, and a MAD extension part of 12 weeks. All subjects will participate in the SAD, MAD, and MAD extension parts, unless they withdraw. End-of-treatment assessments will be performed after 24 weeks of MAD treatment have been completed, i.e. at the Week 25 visit. Subjects will be followed up on adverse events (AEs) and concomitant medications 3 months after the last IMP administration.

An interim analysis will be performed when all subjects in cohort 1 and 2 have completed 12 weeks of MAD treatment. The primary analysis will be performed when all subjects in all cohorts have completed 12 weeks of MAD treatment or discontinued earlier. The final analysis will be performed when all subjects have completed 24 weeks of MAD treatment (12 weeks in the MAD part + 12 weeks in the MAD extension part; Week 25 visit) or discontinued earlier.

As this trial is investigational, there is no defined, expected benefit for subjects who participate in this trial except a better knowledge of their pathology, and the knowledge that they contribute to RNA-targeted therapy for CNM patients carrying MTM1 and DNM2 mutations.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged ≥ 16 years on the date of signing the main Informed Consent Form (ICF).
2. Have a documented mutation in DNM2 or MTM1.
3. Have a symptomatic CNM in the opinion of the investigator, at least mild to moderately affected, i.e. showing clinical symptoms in at least 2 of the relevant 4 domains that will be investigated in this trial (respiratory, muscle strength, muscle function, and dysphagia), and be ambulatory, i.e. being able to walk 10 steps, if needed with support/assisted. If a subject is non-ambulatory but highly functioning in the view of the investigator, he/she may be included following discussion with the sponsor.

5. Have an understanding, ability, and willingness to fully comply with visit frequency, trial procedures and restrictions, including contraceptive requirements.

6. Able to provide written, signed and dated informed consent/assent to participate in the trial. Parental consent (one or both parents) and an assent for subjects < 18 years may be required per local legislation.

Exclusion Criteria:

1. Clinically significant liver disease.
2. Clinically significant renal disease.
3. Presence of significant co-morbidities or conditions other than CNM or clinically significant (CS) findings during screening of medical history, physical examination, laboratory testing, vital signs or ECG recording for which, in the opinion of the investigator and the medical monitor, participation would not be in the best interest of the subject (e.g. compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments (e.g. taking a muscle biopsy).
4. For female subjects of child-bearing potential: pregnant or breastfeeding, or planning to become pregnant during the trial.
5. Current or past abuse of alcohol or recreational/narcotic drugs (with the exception of caffeine and nicotine), which in the investigator's opinion would compromise the subject's safety and/or compliance with the trial procedures.
6. Currently enrolled in any interventional trial or scheduled to participate in such a trial whilst participating in this trial. Subjects are allowed to participate in registry studies.
7. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the IMP or procedures.
8. Intake of any disallowed therapies as noted in Section 5.5 within 12 weeks before the planned first IMP administration.
9. Known or suspected intolerance or hypersensitivity to IMP ingredients or closely-related compounds, or history of a significant allergic reaction to IMP ingredients as determined by the investigator, such as anaphylaxis requiring hospitalization.
10. Legally incapacitated or have limited legal capacity. Lack of mental capacity to fully understand the protocol requirements and complete all study required procedures.

Note: Retesting of subjects should always be discussed with the sponsor and/or medical monitor. Retesting of laboratory values that lead to exclusion will be allowed once using an unscheduled visit during the screening period to assess eligibility. This visit should be at least 2 weeks later than the original screening visit.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Freitag, MD, Study Director — Dynacure; N.C. Voermans, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (8):
- Antwerp University Hospital (UZA), Edegem, Belgium
- Rigshospitalet, Copenhagen Neuromuscular Center, Neurocentret, Copenhagen, Denmark
- Institut de Myologie, Paris, France
- Germany (2):
  - universitätsklinikum Essen, Kinderklinik I, Sozialpädiatrisches Zentrum, Essen
  - Friedrich Baur Institut - Neurologische Klinik LMV, Klinikum Innenstadt, München
- Radboud University Medical Centre, Nijmegen, Netherlands
- United Kingdom (2):
  - MRC centre for Neuromuscular Disease, National Hospital for Neurology and Neurosurgery, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Background info published in Nature on: "Antisense oligonucleotide-mediated Dnm2 knockdown prevents and reverts myotubular myopathy in mice." — https://www.ncbi.nlm.nih.gov/pubmed/28589938

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participant was enrolled in the "Cohort 3 - High Dose" Arm/Group
Groups:
- Cohort 1 - Low Dose: DYN101 in a low dose (1.5 mg/kg weekly IV)
- Cohort 2 - Middle Dose: DYN101 in a middle dose (4.5 mg/kg weekly IV)
- Cohort 3 - High Dose: DYN101 in a high dose (9 mg/kg weekly IV)
Period: Single Ascending Dose (Day 1)
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Started | 6 | 8 | 0
Completed | 6 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Started | 6 | 8 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 8 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 7 | 0
Period: Multiple Ascending Dose Period
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Cohort 3 - High Dose
Started | 6 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Study terminated by Sponsor | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - Low Dose: DYN101 in a low dose (1.5 mg/kg)
- Cohort 2 - Middle Dose: DYN101 in a middle dose (4.5 mg/kg)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Middle Dose | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (16.49) | 37.4 (16.80) | 38.4 (16.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Mutation [Count of Participants; unit: Participants]
  DNM2 | 3 | 5 | 8
  MTM1 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants with drug-related TEAEs during the study period.
Time Frame: Baseline until Study termination, up to 28 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Dose Cohort 1 - Low Dose: DYN101 in a low dose (1.5 mg/kg), single administration
- Single Dose Cohort 2 - Middle Dose: DYN101 in a middle dose (4.5 mg/kg), single administration
- Multiple Dose Cohort 1 - Low Dose: DYN101 in a low dose (1.5 mg/kg), weekly administration
Arm/Group | Single Dose Cohort 1 - Low Dose | Single Dose Cohort 2 - Middle Dose | Multiple Dose Cohort 1 - Low Dose
Number analyzed (Participants) | 6 | 8 | 6
Participants | 1 | 5 | 6

ADVERSE EVENTS:
Time Frame: Baseline until Study termination, up to 28 months
Arm/Group | Single Dose Cohort 1 - Low Dose | Single Dose Cohort 2 - Middle Dose | Multiple Dose Cohort 1 - Low Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose Cohort 1 - Low Dose (N=6) | Single Dose Cohort 2 - Middle Dose (N=8) | Multiple Dose Cohort 1 - Low Dose (N=6)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose Cohort 1 - Low Dose (N=6) | Single Dose Cohort 2 - Middle Dose (N=8) | Multiple Dose Cohort 1 - Low Dose (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 5
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 0
Eye complication associated with device (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 1
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0 | 0
Immunisation reaction (Immune system disorders) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 2
Red blood cells urine positive (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 0
Anxiety (Nervous system disorders) | 1 | 0 | 0
Sleep disorder (Nervous system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Cystatin C increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 3
Total bile acids increased (Investigations) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Investigations) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04033159/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04033159/SAP_001.pdf